CLINICAL TRIAL: NCT04320615
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Safety and Efficacy of Tocilizumab in Patients With Severe COVID-19 Pneumonia
Brief Title: A Study to Evaluate the Safety and Efficacy of Tocilizumab in Patients With Severe COVID-19 Pneumonia
Acronym: COVACTA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA42380; 2020-001154-22 (EudraCT Number)
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Results first posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tocilizumab (TCZ) Arm (Experimental): Participants will receive 1 intravenous (IV) infusion of TCZ, dosed at 8 mg/kg, up to a maximum dose 800 mg. Up to 1 additional dose may be given if clinical symptoms worsen or show no improvement.
  Interventions: Drug: Tocilizumab (TCZ)
- Placebo Arm (Placebo Comparator): Participants will receive 1 IV infusion of placebo matched to TCZ. Up to 1 additional dose may be given if clinical symptoms worsen or show no improvement.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tocilizumab (TCZ) — Participants will receive 1 dose of IV TCZ. 1 additional dose may be given if clinical symptoms worsen or show no improvement.
  Arms: Tocilizumab (TCZ) Arm
Drug: Placebo — Participants will receive 1 dose of IV placebo matched to TCZ. Up to 1 additional dose may be given if clinical symptoms worsen or show no improvement.
  Arms: Placebo Arm

SUMMARY:
This study will evaluate the efficacy, safety, pharmacodynamics, and pharmacokinetics of tocilizumab (TCZ) compared with a matching placebo in combination with standard of care (SOC) in hospitalized patients with severe COVID-19 pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with COVID-19 pneumonia confirmed per WHO criteria (including a positive PCR of any specimen; e.g., respiratory, blood, urine, stool, other bodily fluid) and evidenced by chest X-ray or CT scan
* SPO2 </=93% or PaO2/FiO2 <300 mmHg

Exclusion Criteria:

* Known severe allergic reactions to TCZ or other monoclonal antibodies
* Active tuberculosis (TB) infection
* Suspected active bacterial, fungal, viral, or other infection (besides COVID-19)
* In the opinion of the investigator, progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatments
* Have received oral anti-rejection or immunomodulatory drugs (including TCZ) with the past 3 months
* Participating in other drug clinical trials (participation in COVID-19 anti-viral trials may be permitted if approved by Medical Monitor)
* Pregnant or breastfeeding, or positive pregnancy test in a pre-dose examination
* Treatment with an investigational drug within 5 half-lives or 30 days (whichever is longer) of randomization (investigational COVID-19 antivirals may be permitted if approved by Medial Monitor)
* Any serious medical condition or abnormality of clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 10 x upper limit of normal (ULN) detected within 24 hours at screening (per local lab)
* Absolute neutrophil count (ANC) < 1000/mL at screening (per local lab)
* Platelet count < 50,000/mL at screening (per local lab)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (62):
- United States (23):
  - University of California San Diego, La Jolla, California
  - eStudySite, La Mesa, California
  - David Geffen School of Medicine UCLA, Los Angeles, California
  - Stanford University, Stanford, California
  - Denver Health Medical Center, Denver, Colorado
  - University of Miami Miller School of Medicine, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Ochsner Clinic Foundation, Baton Rouge, Louisiana
  - Baystate Health System, Springfield, Massachusetts
  - Mayo Clinic - PPDS, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Robert Wood Johnson University Hospital/Rutgers, New Brunswick, New Jersey
  - James J Peters Veterans Administration Medical Center - NAVREF, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation; Pulmonary, Allergy & Critical Care Medicine, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Ben Taub General Hospital - HCHD, Houston, Texas
  - Intermountain LDS Hospital, Salt Lake City, Utah
  - Intermountain Medical Group, St. George, Utah
  - Evergreen Health Infectious Disease, Kirkland, Washington
  - Swedish Hospital Medical Center, Seattle, Washington
- Canada (4):
  - Hamilton General Hospital; Pharmacy, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - University Health Network, Toronto, Ontario
  - Clinical Research Institute of Montreal, Montreal, Quebec
- Denmark (4):
  - Rigshospitalet Copenhagen University Hospital, Copenhagen
  - Hvidovre Hospital, Hvidovre
  - Odense Universitetshospital, Odense C
  - Sjællands Universitetshospital, Roskilde, Roskilde
- France (7):
  - Centre Hospitalier Departemental de Vendee, La Roche-sur-Yon
  - Centre Hospitalier et Universitaire de Limoges, Limoges
  - Hôpital de La Croix Rousse, Lyon
  - Hotel Dieu - Nantes, Nantes
  - Hopital de la Pitie Salpetriere, Paris
  - HOPITAL COCHIN university hospital, Paris
  - CHRU de Tours, Pharmacie, Tours
- Germany (4):
  - Universitätsklinikum Köln; Innere Medizin I; Onkologie, Hämatologie, Cologne
  - Universitatsklinikum Dusseldorf, Düsseldorf
  - Medizinische Hochschule Hannover, Hanover
  - LMU Klinikum der Universitat Munchen, München
- Italy (2):
  - Azienda Ospedaliera San Gerardo di Monza, Monza MI, Lombardy
  - Fondazione IRCCS Policlinico San Matteo di Pavia; S.S. Fisiopatologia Respiratoria, Pavia, Lombardy
- Netherlands (4):
  - Amphia Ziekenhuis, Breda
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein
  - Erasmus MC, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Spain (7):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario HM Sanchinarro-CIOCC, Madrid
- United Kingdom (7):
  - Greater Glasgow and Clyde Health Board, Glasgow
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University College Hospital, London
  - Royal Free Hospital, London
  - St George's Clinical Research Facility, London
  - Imperial College London, London
  - North Manchester General Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform https://vivli.org.
  Further details on Roche's criteria for eligible studies are available here: https://vivli.org.
  For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here: (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm

REFERENCES:
- [Derived] Rosas IO, Brau N, Waters M, Go RC, Malhotra A, Hunter BD, Bhagani S, Skiest D, Savic S, Douglas IS, Garcia-Diaz J, Aziz MS, Cooper N, Youngstein T, Sorbo LD, Zerda DJ, Ustianowski A, Gracian AC, Blyth KG, Carratala J, Francois B, Benfield T, Haslem D, Bonfanti P, van der Leest CH, Rohatgi N, Wiese L, Luyt CE, Bauer RN, Cai F, Lee IT, Matharu B, Metcalf L, Wildum S, Graham E, Tsai L, Bao M. Tocilizumab in patients hospitalised with COVID-19 pneumonia: Efficacy, safety, viral clearance, and antibody response from a randomised controlled trial (COVACTA). EClinicalMedicine. 2022 May;47:101409. doi: 10.1016/j.eclinm.2022.101409. Epub 2022 Apr 21. PMID 35475258
- [Derived] Tom J, Bao M, Tsai L, Qamra A, Summers D, Carrasco-Triguero M, McBride J, Rosenberger CM, Lin CJF, Stubbings W, Blyth KG, Carratala J, Francois B, Benfield T, Haslem D, Bonfanti P, van der Leest CH, Rohatgi N, Wiese L, Luyt CE, Kheradmand F, Rosas IO, Cai F. Prognostic and Predictive Biomarkers in Patients With Coronavirus Disease 2019 Treated With Tocilizumab in a Randomized Controlled Trial. Crit Care Med. 2022 Mar 1;50(3):398-409. doi: 10.1097/CCM.0000000000005229. PMID 34612846
- [Derived] Rosas IO, Brau N, Waters M, Go RC, Hunter BD, Bhagani S, Skiest D, Aziz MS, Cooper N, Douglas IS, Savic S, Youngstein T, Del Sorbo L, Cubillo Gracian A, De La Zerda DJ, Ustianowski A, Bao M, Dimonaco S, Graham E, Matharu B, Spotswood H, Tsai L, Malhotra A. Tocilizumab in Hospitalized Patients with Severe Covid-19 Pneumonia. N Engl J Med. 2021 Apr 22;384(16):1503-1516. doi: 10.1056/NEJMoa2028700. Epub 2021 Feb 25. PMID 33631066

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 452 participants were randomized in the study. Of the 452 participants enrolled, 14 were randomized but not dosed and therefore discontinued from the study.
Groups:
- Placebo Modified Intent-to-Treat (mITT) Arm: Participants randomized to the placebo arm who received any amount of study drug. Participants randomized to the placebo arm were to receive 1 IV infusion of placebo matched to TCZ. Up to 1 additional dose could be given if clinical symptoms worsened or showed no improvement.
- Tocilizumab (TCZ) mITT Arm: Participants randomized to the TCZ arm who received any amount of study drug. Participants randomized to the TCZ arm were to receive 1 intravenous (IV) infusion of TCZ, dosed at 8 mg/kg, up to a maximum dose 800 mg. Up to 1 additional dose could be given if clinical symptoms worsened or showed no improvement.
Period: Overall Study
Arm/Group | Placebo Modified Intent-to-Treat (mITT) Arm | Tocilizumab (TCZ) mITT Arm
Started | 144 | 294
Completed | 96 | 190
Not Completed | 48 | 104
Not completed — Withdrawal by Subject | 4 | 10
Not completed — Physician Decision | 2 | 0
Not completed — Other | 2 | 0
Not completed — Lost to Follow-up | 5 | 23
Not completed — Death | 35 | 71

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Modified Intent-to-Treat (mITT) Arm | Tocilizumab (TCZ) mITT Arm | Total
Number analyzed (Participants) | 144 | 294 | 438
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.6 (13.7) | 60.9 (14.6) | 60.8 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 89 | 132
  Male | 101 | 205 | 306
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 94 | 141
  Not Hispanic or Latino | 86 | 181 | 267
  Unknown or Not Reported | 11 | 19 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 8 | 13
  Asian | 10 | 28 | 38
  Native Hawaiian or Other Pacific Islander | 5 | 3 | 8
  Black or African American | 26 | 40 | 66
  White | 76 | 176 | 252
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 21 | 39 | 60

OUTCOME MEASURES:

1. Primary Outcome: Clinical Status Assessed Using a 7-Category Ordinal Scale at Day 28 (Week 4)
Description: Clinical status was assessed using a 7-category ordinal scale:
  1. - Discharged (or "ready for discharge")
  2. - Non- intensive care unit (ICU) hospital ward (or "ready for hospital ward") not requiring supplemental oxygen
  3. - Non-ICU hospital ward (or "ready for hospital ward") requiring supplemental oxygen
  4. - ICU or non-ICU hospital ward, requiring non-invasive ventilation or high-flow oxygen
  5. - ICU, requiring intubation and mechanical ventilation
  6. - ICU, requiring extracorporeal membrane oxygenation (ECMO) or mechanical ventilation and additional organ support
  7. - Death
Time Frame: Day 28
Population: mITT population: Defined as all randomized participants who received any amount of study medication, with participants grouped according to the treatment assigned at randomization.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab (TCZ) mITT Arm | Placebo Modified Intent-to-Treat (mITT) Arm
Number analyzed (Participants) | 294 | 144
Percentage of Participants
  1 | 56.5 | 49.3
  2 | 2.0 | 5.6
  3 | 4.8 | 2.8
  4 | 2.0 | 6.9
  5 | 8.8 | 9.7
  6 | 6.1 | 6.3
  7 | 19.7 | 19.4
Statistical Analysis 1: Comparison: Tocilizumab (TCZ) mITT Arm vs Placebo Modified Intent-to-Treat (mITT) Arm; Test type: Other; p = 0.3600, Van Elteren Test; Median Difference (Final Values) = -1.0, 95% CI 2-sided [-2.5 to 0.0]

2. Secondary Outcome: Time to Clinical Improvement (TTCI), Defined as a National Early Warning Score 2 (NEWS2) of </= 2 Maintained for 24 Hours
Description: Defined as time from first dose of study drug to at least two NEWS2 assessments with a score of <=2 covering a span of at least 21.5 hours, with a maximum of 26.5 hours between the first and last of these assessments and no assessments with a score >2 in between. If one of the components of the NEWS2 score was missing at a particular time point, then the NEWS2 score was not calculated. Participants who died were censored at Day 28.
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tocilizumab (TCZ) mITT Arm | Placebo Modified Intent-to-Treat (mITT) Arm
Number analyzed (Participants) | 294 | 144
Days | NA [NA to NA] — NA = Value not estimable (NE) due to an insufficient number of events. | NA [NA to NA] — NA = Value not estimable (NE) due to an insufficient number of events.
Statistical Analysis 1: Comparison: Tocilizumab (TCZ) mITT Arm vs Placebo Modified Intent-to-Treat (mITT) Arm; Test type: Other; p = 0.0443, Log Rank; Hazard Ratio (HR) = 1.448, 95% CI 2-sided [1.01 to 2.08]

3. Secondary Outcome: Time to Improvement of at Least 2 Categories Relative to Baseline on a 7-Category Ordinal Scale of Clinical Status
Description: Time to improvement for this outcome measure was defined as the days from the first dose of study drug to when at least a 2-category improvement in clinical status (based on a 7-category ordinal scale) is observed. Participants who died were censored at Day 28.
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tocilizumab (TCZ) mITT Arm | Placebo Modified Intent-to-Treat (mITT) Arm
Number analyzed (Participants) | 294 | 144
Days | 14.0 [12.0 to 17.0] | 18.0 [15.0 to 28.0]
Statistical Analysis 1: Comparison: Tocilizumab (TCZ) mITT Arm vs Placebo Modified Intent-to-Treat (mITT) Arm; Test type: Other; p = 0.0820, Log Rank; Hazard Ratio (HR) = 1.263, 95% CI 2-sided [0.97 to 1.64]

4. Secondary Outcome: Time to Hospital Discharge or "Ready for Discharge"
Description: Time to Hospital Discharge was defined as the time from the first dose of study drug to hospital discharge or "ready for discharge" (normal body temperature and respiratory rate, and stable oxygen saturation on ambient air or </=2L supplemental oxygen) Participants who died were censored at Day 28.
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tocilizumab (TCZ) mITT Arm | Placebo Modified Intent-to-Treat (mITT) Arm
Number analyzed (Participants) | 294 | 144
Days | 20.0 [17.0 to 27.0] | 28.0 [20.0 to NA] — NA = Value not estimable (NE) due to an insufficient number of events.
Statistical Analysis 1: Comparison: Tocilizumab (TCZ) mITT Arm vs Placebo Modified Intent-to-Treat (mITT) Arm; Test type: Other; p = 0.0370, Log Rank; Hazard Ratio (HR) = 1.350, 95% CI 2-sided [1.02 to 1.79]

5. Secondary Outcome: Incidence of Mechanical Ventilation by Day 28
Description: Participants who died by Day 28 were assumed to have required mechanical ventilation.
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- TCZ - No Mechanical Ventilation at Baseline: Participants randomized to the TCZ arm who received any amount of study drug and were not on mechanical ventilation at baseline. Participants randomized to the TCZ arm were to receive 1 intravenous (IV) infusion of TCZ, dosed at 8 mg/kg, up to a maximum dose 800 mg. Up to 1 additional dose could be given if clinical symptoms worsened or showed no improvement.
- Placebo - No Mechanical Ventilation at Baseline: Participants randomized to the placebo arm who received any amount of study drug and were not on mechanical ventilation at baseline. Participants randomized to the placebo arm were to receive 1 IV infusion of placebo matched to TCZ. Up to 1 additional dose could be given if clinical symptoms worsened or showed no improvement.
Arm/Group | Tocilizumab (TCZ) mITT Arm | Placebo Modified Intent-to-Treat (mITT) Arm | TCZ - No Mechanical Ventilation at Baseline | Placebo - No Mechanical Ventilation at Baseline
Number analyzed (Participants) | 294 | 144 | 183 | 90
Percentage of Participants | 54.4 [48.7 to 60.1] | 60.4 [52.4 to 68.4] | 27.9 [21.4 to 34.4] | 36.7 [26.7 to 46.6]
Statistical Analysis 1: Comparison: Tocilizumab (TCZ) mITT Arm vs Placebo Modified Intent-to-Treat (mITT) Arm; Test type: Other; p = 0.0996, Cochran-Mantel-Haenszel; Weighted % difference = -6.2, 95% CI 2-sided [-13.8 to 1.4]
Statistical Analysis 2: Comparison: TCZ - No Mechanical Ventilation at Baseline vs Placebo - No Mechanical Ventilation at Baseline; Test type: Other; p = 0.1355, Cochran-Mantel-Haenszel; Weighted % difference = -8.9, 95% CI 2-sided [-20.7 to 3.0]

6. Secondary Outcome: Ventilator-Free Days to Day 28
Description: Participants who died by Day 28 were assigned 0 ventilator-free days.
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tocilizumab (TCZ) mITT Arm | Placebo Modified Intent-to-Treat (mITT) Arm
Number analyzed (Participants) | 294 | 144
Days | 22.0 [18.0 to 28.0] | 16.5 [11.0 to 26.0]
Statistical Analysis 1: Comparison: Tocilizumab (TCZ) mITT Arm vs Placebo Modified Intent-to-Treat (mITT) Arm; Test type: Other; p = 0.3202, Van Elteren test; Median Difference (Final Values) = 5.5, 95% CI 2-sided [-2.8 to 13.0]

7. Secondary Outcome: Incidence of Intensive Care Unit (ICU) Stay by Day 28 (Week 4)
Description: Participants who died by Day 28 were assumed to have required an ICU stay.
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- TCZ - Not in ICU at Baseline: Participants randomized to the TCZ arm who received any amount of study drug and were not in the ICU at baseline. Participants randomized to the TCZ arm were to receive 1 intravenous (IV) infusion of TCZ, dosed at 8 mg/kg, up to a maximum dose 800 mg. Up to 1 additional dose could be given if clinical symptoms worsened or showed no improvement.
- Placebo - Not in ICU at Baseline: Participants randomized to the placebo arm who received any amount of study drug and were not in the ICU at baseline. Participants randomized to the placebo arm were to receive 1 IV infusion of placebo matched to TCZ. Up to 1 additional dose could be given if clinical symptoms worsened or showed no improvement.
Arm/Group | Tocilizumab (TCZ) mITT Arm | Placebo Modified Intent-to-Treat (mITT) Arm | TCZ - Not in ICU at Baseline | Placebo - Not in ICU at Baseline
Number analyzed (Participants) | 294 | 144 | 127 | 64
Percentage of Participants | 66.0 [60.6 to 71.4] | 71.5 [64.2 to 78.9] | 21.3 [14.1 to 28.4] | 35.9 [24.2 to 47.7]
Statistical Analysis 1: Comparison: Tocilizumab (TCZ) mITT Arm vs Placebo Modified Intent-to-Treat (mITT) Arm; Test type: Other; p = 0.1514, Cochran-Mantel-Haenszel; Weighted % difference = -5.7, 95% CI 2-sided [-13.7 to 2.2]
Statistical Analysis 2: Comparison: TCZ - Not in ICU at Baseline vs Placebo - Not in ICU at Baseline; Test type: Other; p = 0.0290, Cochran-Mantel-Haenszel; Weighted % difference = -14.8, 95% CI 2-sided [-28.6 to -1.0]

8. Secondary Outcome: Duration of ICU Stay to Day 28 (Week 4)
Description: Participants who died by Day 28 were assigned a duration from the first dose of study drug to Day 28 at hour 23:59:59.
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tocilizumab (TCZ) mITT Arm | Placebo Modified Intent-to-Treat (mITT) Arm
Number analyzed (Participants) | 294 | 144
Days | 9.8 [7.0 to 15.7] | 15.5 [8.7 to 25.5]
Statistical Analysis 1: Comparison: Tocilizumab (TCZ) mITT Arm vs Placebo Modified Intent-to-Treat (mITT) Arm; Test type: Other; p = 0.0454, Van Elteren test; Median Difference (Final Values) = -5.8, 95% CI 2-sided [-15.0 to 2.9]

9. Secondary Outcome: Clinical Status Assessed Using a 7-Category Ordinal Scale at Day 14
Description: as for outcome 1
Time Frame: Day 14
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab (TCZ) mITT Arm | Placebo Modified Intent-to-Treat (mITT) Arm
Number analyzed (Participants) | 294 | 144
Percentage of participants
  1 | 39.8 | 29.9
  2 | 6.1 | 4.9
  3 | 6.5 | 11.1
  4 | 7.1 | 7.6
  5 | 14.6 | 16.0
  6 | 12.6 | 17.4
  7 | 13.3 | 13.2
Statistical Analysis 1: Comparison: Tocilizumab (TCZ) mITT Arm vs Placebo Modified Intent-to-Treat (mITT) Arm; Test type: Other; p = 0.0548, Van Elteren test; Median Difference (Final Values) = -1.0, 95% CI 2-sided [-2.0 to 0.5]

10. Secondary Outcome: Time to Clinical Failure to Day 28 (Week 4)
Description: Time to clinical failure was defined as the number of days from the first dose of study drug to the first occurrence on study of death, mechanical ventilation, ICU admission, or study withdrawal prior to discharge, whichever occurs first.
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tocilizumab (TCZ) mITT Arm | Placebo Modified Intent-to-Treat (mITT) Arm
Number analyzed (Participants) | 294 | 144
Days | NA [NA to NA] — NA = Value not estimable (NE) due to an insufficient number of events. | NA [21.0 to NA] — NA = Value not estimable (NE) due to an insufficient number of events.
Statistical Analysis 1: Comparison: Tocilizumab (TCZ) mITT Arm vs Placebo Modified Intent-to-Treat (mITT) Arm; Test type: Other; p = 0.1627, Log Rank; Hazard Ratio (HR) = 0.790, 95% CI 2-sided [0.57 to 1.10]

11. Secondary Outcome: Mortality Rate at Day 28 (Week 4)
Time Frame: Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tocilizumab (TCZ) mITT Arm | Placebo Modified Intent-to-Treat (mITT) Arm
Number analyzed (Participants) | 294 | 144
Percentage of Participants | 19.7 [15.2 to 24.3] | 19.4 [13.0 to 25.9]
Statistical Analysis 1: Comparison: Tocilizumab (TCZ) mITT Arm vs Placebo Modified Intent-to-Treat (mITT) Arm; Test type: Other; p = 0.9410, Cochran-Mantel-Haenszel; Weighted % difference = 0.3, 95% CI 2-sided [-7.6 to 8.2]

12. Secondary Outcome: Time to Recovery to Day 28 (Week 4)
Description: Time to recovery was defined as the number of days from the first dose of study drug to hospital discharge or "ready for discharge" (normal body temperature and respiratory rate, and stable oxygen saturation on ambient air or </= 2L supplemental oxygen) or non-ICU hospital ward or "ready for hospital ward" not requiring supplemental oxygen. Participants who died were censored at Day 28.
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tocilizumab (TCZ) mITT Arm | Placebo Modified Intent-to-Treat (mITT) Arm
Number analyzed (Participants) | 294 | 144
Days | 16.0 [12.0 to 21.0] | 24.0 [18.0 to NA] — NA = Value not estimable (NE) due to an insufficient number of events.
Statistical Analysis 1: Comparison: Tocilizumab (TCZ) mITT Arm vs Placebo Modified Intent-to-Treat (mITT) Arm; Test type: Other; p = 0.0528, Log Rank; Hazard Ratio (HR) = 1.307, 95% CI 2-sided [1.00 to 1.72]

13. Secondary Outcome: Duration of Supplemental Oxygen to Day 28 (Week 4)
Description: Participants who died by Day 28 were assigned a duration of 28 days of supplemental oxygen.
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tocilizumab (TCZ) mITT Arm | Placebo Modified Intent-to-Treat (mITT) Arm
Number analyzed (Participants) | 294 | 144
Days | 26.5 [19.0 to 28.0] | 28.0 [26.0 to 28.0]
Statistical Analysis 1: Comparison: Tocilizumab (TCZ) mITT Arm vs Placebo Modified Intent-to-Treat (mITT) Arm; Test type: Other; p = 0.0477, Van Elteren test; Median Difference (Final Values) = -1.5, 95% CI 2-sided [-9.0 to 0.5]

ADVERSE EVENTS:
Time Frame: 60 days
Description: The safety-evaluable population consisted of all participants who received any amount of study medication. Participants are grouped according to the treatment first received rather than the treatment assigned at randomization.
Groups:
- Placebo Arm (Safety-Evaluable Population); Tocilizumab (TCZ) Arm (Safety-Evaluable Population): The safety-evaluable population consisted of all participants who received any amount of study medication. Participants are grouped according to the treatment first received rather than the treatment assigned at randomization.
Arm/Group | Placebo Arm (Safety-Evaluable Population) | Tocilizumab (TCZ) Arm (Safety-Evaluable Population)
All-Cause Mortality (participants affected / at risk) | 36/143 | 72/295
Serious Adverse Events (participants affected / at risk) | 64/143 | 116/295
Other Adverse Events (participants affected / at risk) | 29/143 | 83/295
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Arm (Safety-Evaluable Population) (N=143) | Tocilizumab (TCZ) Arm (Safety-Evaluable Population) (N=295)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (3)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 5 (6) | 4 (4)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 2 (2)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 2 (2) | 2 (2)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal hernia perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 2 (2)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 5 (5)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 3 (3) | 3 (3)
Bacterial sepsis (Infections and infestations) | 0 (0) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 14 (14)
COVID-19 pneumonia (Infections and infestations) | 20 (20) | 36 (36)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus hepatitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (5) | 7 (8)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 6 (6)
Pneumonia escherichia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 3 (3)
Septic shock (Infections and infestations) | 7 (8) | 7 (7)
Staphylococcal infection (Infections and infestations) | 1 (1) | 1 (1)
Stenotrophomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transfusion-related acute lung injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Citrobacter test positive (Investigations) | 0 (0) | 1 (1)
Enterococcus test positive (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic transformation stroke (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 10 (10)
Renal failure (Renal and urinary disorders) | 2 (2) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Arm (Safety-Evaluable Population) (N=143) | Tocilizumab (TCZ) Arm (Safety-Evaluable Population) (N=295)
Anaemia (Blood and lymphatic system disorders) | 10 (10) | 17 (17)
Constipation (Gastrointestinal disorders) | 8 (8) | 18 (18)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 18 (18)
Pneumonia (Infections and infestations) | 8 (12) | 10 (10)
Urinary tract infection (Infections and infestations) | 5 (6) | 22 (22)
Hypertension (Vascular disorders) | 3 (4) | 20 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/15/NCT04320615/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/15/NCT04320615/SAP_001.pdf